CLINICAL TRIAL: NCT07360808
Title: Safety and Efficacy of Autologous Adipose-Derived Regenerative Cells (ADRCs) for Improving Hand Dysfunction in Systemic Sclerosis: A Prospective, Randomized, Multicenter Superiority Trial
Brief Title: Safety and Efficacy of Adipose-Derived Regenerative Cells (ADRCs) for Improving Hand Dysfunction in Systemic Sclerosis
Acronym: AEGIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cytori Therapeutics (Industry)
Collaborators: Huashan Hospital (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEGIS
Record Dates: First submitted 2025-11-21; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Systemic Sclerosis (SSc); Hand Dysfunction
Keywords: Adipose-Derived Regenerative Cells (ADRCs); Systemic Sclerosis; Hand Function; Raynaud Condition
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADRCs group (Experimental)
  Interventions: Device: Autologous ADRCs injection Combined with Standard Therapy
- Standard Treatment group (Other)
  Interventions: Drug: Standard Treatment group

INTERVENTIONS:
Device: Autologous ADRCs injection Combined with Standard Therapy — Liposuction harvests ≥180 mL adipose tissue from the subject's abdomen/thighs or other suitable sites. Tissue is cleaned/separated via Celution 800/GP to obtain ADRCs, whose total volume is adjusted to 10 mL with lactated Ringer's solution.
  On treatment day, single retrograde injection is given to each finger of both hands (1 mL total per finger).
  Both thumbs: Injection sites on both sides of metacarpophalangeal joint. Insert 25G sharp needle from joint to thumb's distal end; switch to 25G blunt needle for subcutaneous retrograde injection (distal→proximal). 0.5 mL per side, total 1 mL.
  Other fingers: Injection sites on both sides of proximal interphalangeal joint (palmar-dorsal skin junction). Insert 25G sharp needle toward finger's proximal/distal ends; switch to 25G blunt needle for injection (distal→joint, proximal→joint). 0.25 mL per direction per side (0.5 mL/side), total 1 mL ADRCs per finger.
  Arms: ADRCs group
Drug: Standard Treatment group — The standard treatment refers to the routine treatment plan formulated by researchers for subjects in accordance with the "Diagnosis and Treatment Standards for Systemic Sclerosis" and based on the specific conditions of the patients.
  Arms: Standard Treatment group

SUMMARY:
This prospective, randomized, blinded, multicenter clinical study aims to evaluate the safety and efficacy of autologous adipose-derived regenerative cells (ADRCs) in improving hand dysfunction in patients with systemic sclerosis (SSc). The study plans to enroll 48 eligible patients, randomly assigned to two groups. The experimental group will receive ADRCs, prepared from the Celution system, which is injected into specific sites on each finger of both hands. The control group will receive standard care according to established treatment guidelines. The primary endpoint is the change from baseline in the Cochin Hand Function Scale (CHFS) score at 24 weeks. Secondary endpoints include assessments of skin thickness, Raynaud phenomenon, hand strength, quality of life, pain, and other measures at various time points. Safety and device performance will be monitored throughout the study. This investigation seeks to explore a new potential therapeutic direction for managing hand dysfunction in systemic sclerosis.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) often preferentially affects the hands, leading to skin thickening, limited mobility, pain, and even digital ulcers, severely impairing hand function and quality of life in patients. This prospective, randomized, multicenter, superiority-designed clinical study aims to evaluate the safety and efficacy of autologous adipose-derived regenerative cells (ADRCs) prepared using the Celution 800/GP System and the Celution 805 for improving hand dysfunction in patients with systemic sclerosis.

The study plans to enroll 48 eligible patients, randomly assigned to two groups. For the ADRCs group, at least 180 mL of autologous adipose tissue was obtained via liposuction. The Celution 800/GP system and Celution 805 were used to wash, separate, and enrich the ADRCs. These were then adjusted to a volume of 10 mL using Lactated Ringer's solution (divided into 10 syringes of 1 mL each) and injected into specific sites on each finger of both hands (both sides of the metacarpophalangeal joint of the thumb and both sides of the proximal interphalangeal joints of the other fingers). The control group received standard treatment guided by the "Diagnosis and Treatment Guidelines for Systemic Sclerosis." Patients were randomly assigned to the two groups in a 1:1 ratio. Participants were followed up multiple times within 4 weeks, 12 weeks, and 24 weeks post-procedure.

The primary endpoint was the change from baseline in the Cochin Hand Function Scale (CHFS) score at 24 weeks. Secondary endpoints included changes from baseline in the CHFS score at 4 and 12 weeks; the modified Rodnan skin score at 4, 12, and 24 weeks; Raynaud's Condition Score; Kapandji score; hand grip strength/pinch strength; Systemic Sclerosis Health Assessment Questionnaire (SHAQ) score; pain Visual Analogue Scale (VAS) score; and digital ulcer clinical assessment scale score at the respective timepoints. Additionally, changes from baseline in hand skin ultrasound examination and nailfold capillaroscopy results at 24 weeks were assessed. Performance evaluation of the Celution800/GP system and Celution805, monitoring of safety indicators, and device deficiencies were also included.

Statistical analysis followed standard principles using SAS software (version 9.4). Efficacy analyses were performed using data from both the Full Analysis Set and the Per-Protocol Set, while safety analyses used the Safety Analysis Set.

This study focuses on the safety and efficacy of autologous ADRCs in treating hand dysfunction in systemic sclerosis, offering a new direction for improving hand dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old (inclusive), gender not restricted;
2. According to the 2013 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) systemic sclerosis (SSc) diagnostic criteria, diagnosed as diffuse cutaneous type or localized cutaneous type;
3. Thickened hand skin, modified Rodnan skin score ≥ 8 points and ≤ 35 points;
4. Cochin Hand Function Scale (CHFS) ≥ 20 (total score 90), with or without skin ulcers;
5. Capable of safely undergoing liposuction to obtain sufficient adipose tissue (the preferred fat extraction sites are the abdomen, followed by the lateral abdomen, inner and outer thighs, posterior thighs, and anterior thighs; multiple sites can be selected for liposuction to obtain sufficient adipose tissue);
6. Voluntary participation in this clinical trial and signing the informed consent form by the subject.

Exclusion Criteria:

1. Subject's body mass index (BMI) < 17 kg/m^2;
2. Hand skin lesions are in the atrophic stage, and the investigator determines that they are not suitable for hand drug injection;
3. Any finger contracture or injection site ulcer that makes it unsafe to complete the injection;
4. Any proximal to distal interphalangeal joint amputation of any finger, or amputation of more than one finger;
5. Concurrent other rheumatic immune diseases, such as RA, SLE, dermatomyositis, etc. (existing rheumatic immune diseases that do not affect the safety and efficacy evaluation of the hand and do not affect the safety of the hand and efficacy evaluation, excluding Sjögren's syndrome);
6. Active infectious diseases or patients who have used antibiotics within 3 months before the screening visit due to active infectious diseases;
7. Patients with unstable systemic sclerosis who have received cell therapy before the screening visit;
8. Patients who have undergone chemotherapy or resection of malignant cancer within 5 years before the screening visit;
9. Abnormal tumor markers detected during the screening period, and the investigator determines that there is a tumor risk;
10. Patients who have received CD20 monoclonal antibody treatment within 1 year before the screening visit, or have used other biologic drugs or taken small molecule targeted drugs within 3 months before the screening visit (excluding those who have maintained a stable dose of ≥ 3 months at the time of enrollment for systemic sclerosis treatment);
11. Have received hand cell injection therapy before, or are intolerant to cell therapy, or have received systemic cell injection therapy within 6 months before the screening visit;
12. Patients with positive human immunodeficiency virus antibody (anti-HIV-Ab) test results, active syphilis, active hepatitis C (HCV-RNA positive, and hepatitis C antibody positive), hepatitis B (HBsAg positive and HBV-DNA positive) during the screening period;
13. There is evidence indicating that the subject currently has possible safety-related diseases in the digestive system, urinary system, cardiovascular system, hematological system, nervous system, mental state, and metabolism, such as poorly controlled diabetes, poorly controlled hypertension, etc.;
14. Any of the following laboratory test results during the screening period: ① Abnormal blood routine: hemoglobin < 80 g/L; white blood cell count < 3.0 × 10^9/L; absolute neutrophil count < 1.2 × 10^9/L; platelet count < 100 × 10^9/L; ② Abnormal liver and kidney function: aspartate transaminase (AST), alanine aminotransferase (ALT), activated partial thromboplastin time (APTT) prolonged > 1.5 times the upper limit of the reference value; ③ Coagulation dysfunction: prothrombin time (PT) and partial thromboplastin time (APTT) prolonged > 1.8 times the upper limit of the reference value, or international normalized ratio (INR) > 2;
15. Allergic to any component of human albumin, anesthetic drugs, or human adipose-derived mesenchymal stem cell injection solution, or the investigator determines that the subject is not suitable for enrollment due to a severe allergy history;
16. Patients whose screening visit is within 3 months before the general anesthesia surgery planned during the study period;
17. Patients who have participated in other clinical studies within 3 months before the screening visit, or are currently participating in other clinical studies;
18. Pregnant women, lactating women, those with positive pregnancy test results, or those who do not agree to use effective contraceptive measures during the study period and within 6 months after the trial;
19. Patients judged by the investigator to be unsuitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cochin Hand Function Scale (CHFS) Score from baseline | Screening period (-30 to -1 day), 24 weeks post-treatment (±7 days)
  The assessment tool comprises 18 items across five dimensions: kitchen skills (8 items), dressing (2 items), personal hygiene (2 items), work competency (2 items), and other daily living activities (4 items). Each item is scored on a 0-5 scale, where "no difficulty" scores 0 and "inability" scores 5. The total score ranges from 0 to 90 points, with higher scores indicating more severe hand function impairment.

SECONDARY OUTCOMES:
Change in Cochin Hand Function Scale (CHFS) Score from baseline | Screening period (-30 to -1 day), 4 weeks (±3 days) and 12 weeks (±7 days) post-treatment
  The assessment tool comprises 18 items across five dimensions: kitchen skills (8 items), dressing (2 items), personal hygiene (2 items), work competency (2 items), and other daily living activities (4 items). Each item is scored on a 0-5 scale, where "no difficulty" scores 0 and "inability" scores 5. The total score ranges from 0 to 90 points, with higher scores indicating more severe hand function impairment.
Change in modified Rodnan Skin Score (mRSS) from baseline | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
  The researchers evaluated the modified Rodnan Skin Score (mRSS), which assesses skin thickness across 17 different body areas. Each area is rated on a 0-3 scale, with a total score of 51. Higher scores indicate more severe skin fibrosis.
Change in Raynaud Condition Score (RCS) from baseline | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
  The evaluation was conducted by the subjects. The Raynaud Condition Score (RCS) assesses the degree of sensory difficulty in the patient's hands. The RCS is a self-assessment of daily Raynaud Phenomenon (RP) activity, including the daily cumulative frequency, duration, severity, and impact of RP episodes. It is evaluated using a 0-10 rating scale via standardized scoring rules. Subjects record the number of RP episodes per day and the duration of each episode (in minutes), and complete the Raynaud Condition Score (RCS). The researchers calculate and record the average score of the subjects' Raynaud values.
Change in Kapandji Score from baseline | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
  The evaluation is conducted by the researchers. Based on the position where the thumb tip can be reached when each finger is fully extended, the following 10 areas are assessed: ① the radial side of the middle joint of the index finger, ② the radial side of the distal joint of the index finger, ③ the tip of the index finger, ④ the tip of the middle finger, ⑤ the tip of the ring finger, ⑥ the tip of the little finger, ⑦ the radial side of the distal interphalangeal joint of the little finger, ⑧ the proximal end of the little finger (near the nail), ⑨ the radial side of the metacarpophalangeal joint of the little finger, ⑩ the distal palmar line. These 10 areas represent scores of 1 to 10 respectively.
Change in Hand Grip Strength from baseline | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
  The evaluation is conducted by the researchers. Subject position: Sit quietly in a upright position, with the shoulder joint at 0 degrees, the elbow at 90 degrees, the upper arm flat against the chest, the forearm in a neutral position, and the wrist at 30 degrees of extension. Instruct the subjects to exert their maximum effort to measure the grip strength of both hands. Repeat the measurement three times, with a rest period for the subjects between each measurement to eliminate test fatigue. Take the average of the three test results as the final test result.
Change in Hand Pinch Strength from baseline | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
  The evaluation is conducted by the researchers. Subject position: Sit quietly in a upright position, with the shoulder joint at 0 degrees, the elbow at 90 degrees, the upper arm flat against the chest, the forearm in a neutral position, and the wrist at 30 degrees of extension. Instruct the subjects to exert their maximum effort to measure the pinch force of both hands. Repeat the measurement three times, with a rest period for the subjects between each measurement to eliminate test fatigue. Take the average of the three test results as the final test result.
Change in Hand Skin Ultrasound from baseline | Screening period (-30 to -1 day) and 24 weeks (±7 days) post-treatment
  The evaluation was conducted by the researchers. The thickness of the skin on the hands was measured using ultrasound.
Change in Nailfold Microcirculation from baseline | Screening period (-30 to -1 day) and 24 weeks (±7 days) post-treatment
  The evaluation was conducted by the researchers. The nailfold microcirculation examination assesses the severity of microvascular lesions in the fingers of both hands (excluding the thumbs).
Change in Systemic Sclerosis Health Assessment Questionnaire (SHAQ) Score from baseline | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
  The evaluation is conducted by the subjects. SHAQ consists of two parts: ① The standard HAQ section (8 types of daily activities), which assesses the ability to perform daily activities and the tools and assistance required for completing daily activities; ② Specific additional questions for systemic sclerosis include 5 visual analogue scales (VAS), covering the impact of Raynaud's phenomenon; gastrointestinal symptoms; respiratory system symptoms; skin tightness; and overall assessment of disease severity.
Change in Pain Visual Analogue Scale (VAS) Score from baseline | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
  The evaluation is conducted by the subjects.The evaluation is conducted by the subjects. The subjects mark the corresponding position on this line to represent the intensity of the pain they experienced at that moment. The distance from the starting point to the marking point is measured to obtain the pain score. The higher the score, the more intense the pain.
Change in Digital Ulcer Clinical Assessment Scale Score (HDISS-DU) from baseline | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
  The evaluation was conducted by blind assessors. The impact of scleroderma-related fingertip ulcers on hand function was assessed using the HDISS-DU scale. Twenty-four questions were posed over a 7-day observation period, with answer scores ranging from 1 to 6. A score of 1 indicated "can, without difficulty", while a score of 6 indicated "cannot". A score of 5 indicated "almost impossible" or "can only be completed with the unaffected hand that is not ulcerated".
Equipment performance evaluation | 0 day
  Incidence of breakage of connecting components, loosening and falling off of components, and electric leakage of the control system in the Celution800/GP system (%)

OTHER OUTCOMES:
Vital signs: body temperature | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Vital signs: respiration | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Vital signs: pulse | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Vital signs: blood pressure | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
  systolic and diastolic
Laboratory tests: Red Blood Cell (RBC) Count | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: White Blood Cell (WBC) Count | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Platelets (PLT) Count | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Hemoglobin (HB) Concentration | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Neutrophil (NEUT) Percentage | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Urinary Protein (PRO) | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
  Qualitative result (＋/-)
Laboratory tests: Urinary Glucose (GLU) | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
  Qualitative result (＋/-)
Laboratory tests: Urinary White Blood Cells (WBC) Count | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Urinary Red Blood Cells (RBC) Count | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Aspartate Aminotransferase (AST) | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Alanine Aminotransferase (ALT) | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Creatinine (Cr) | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Blood Urea Nitrogen (BUN)/Urea | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Activated Partial Thromboplastin Time (APTT) | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Prothrombin Time (PT) | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Fibrinogen (FIB) | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Thrombin Time (TT) | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: Fibrin (Fibrinogen) Degradation Products (FDP) | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Laboratory tests: D-Dimer (D-D) | Screening period (-30 to -1 day), 4 weeks (±3 days), 12 weeks (±7 days) and 24 weeks (±7 days) post-treatment
Incidence of Adverse Events, Incidence of Serious Adverse Events | From Day 0 through the completion of follow-up.Each individual participant will undergo a 24 weeks follow-up period, and it is anticipated that all follow-up assessments will be completed by December 31, 2027.
Device defects: Incidence Rate of Medical Device Malfunctions | 0 day

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - NanFang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Huashan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No